CLINICAL TRIAL: NCT01526213
Title: Do Furanocoumarins Mediate the Fexofenadine-grapefruit Juice Interaction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB 09-0788
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2012-12

CONDITIONS: Food-drug Interaction
MeSH Terms: interventions — fexofenadine; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1: Water, GFJ, FC-free GFJ (Other): This randomized, open-label, single-dose, 3-way crossover study in healthy volunteers will be conducted in the CTRC. Once subjects are identified as eligible to participate, based on their screening evaluation and according to inclusion/exclusion criteria, they will undergo 3 phases. By randomized crossover design, the subject will receive fexofenadine with water, grapefruit juice (GFJ), or furanocoumarin (FC)-free grapefruit juice.
  Interventions: Drug: Fexofenadine
- Sequence 2: Water, FC-free GFJ, GFJ (Other): This randomized, open-label, single-dose, 3-way crossover study in healthy volunteers will be conducted in the CTRC. Once subjects are identified as eligible to participate, based on their screening evaluation and according to inclusion/exclusion criteria, they will undergo 3 phases. By randomized crossover design, the subject will receive fexofenadine with water, grapefruit juice (GFJ), or furanocoumarin (FC)-free grapefruit juice.
  Interventions: Drug: Fexofenadine
- Sequence 3: GFJ, FC-free GFJ, Water (Other): This randomized, open-label, single-dose, 3-way crossover study in healthy volunteers will be conducted in the CTRC. Once subjects are identified as eligible to participate, based on their screening evaluation and according to inclusion/exclusion criteria, they will undergo 3 phases. By randomized crossover design, the subject will receive fexofenadine with water, grapefruit juice (GFJ), or furanocoumarin (FC)-free grapefruit juice.
  Interventions: Drug: Fexofenadine
- Sequence 4: GFJ, Water, FC-free GFJ (Other): This randomized, open-label, single-dose, 3-way crossover study in healthy volunteers will be conducted in the CTRC. Once subjects are identified as eligible to participate, based on their screening evaluation and according to inclusion/exclusion criteria, they will undergo 3 phases. By randomized crossover design, the subject will receive fexofenadine with water, grapefruit juice (GFJ), or furanocoumarin (FC)-free grapefruit juice.
  Interventions: Drug: Fexofenadine
- Sequence 5: FC-free GFJ, GFJ, Water (Other): This randomized, open-label, single-dose, 3-way crossover study in healthy volunteers will be conducted in the CTRC. Once subjects are identified as eligible to participate, based on their screening evaluation and according to inclusion/exclusion criteria, they will undergo 3 phases. By randomized crossover design, the subject will receive fexofenadine with water, grapefruit juice (GFJ), or furanocoumarin (FC)-free grapefruit juice.
  Interventions: Drug: Fexofenadine
- Sequence 6: FC-free GFJ, Water, GFJ (Other): This randomized, open-label, single-dose, 3-way crossover study in healthy volunteers will be conducted in the CTRC. Once subjects are identified as eligible to participate, based on their screening evaluation and according to inclusion/exclusion criteria, they will undergo 3 phases. By randomized crossover design, the subject will receive fexofenadine with water, grapefruit juice (GFJ), or furanocoumarin (FC)-free grapefruit juice.
  Interventions: Drug: Fexofenadine

INTERVENTIONS:
Drug: Fexofenadine — This randomized, open-label, single-dose, 3-way crossover study in healthy volunteers will be conducted in the CTRC. Once subjects are identified as eligible to participate, based on their screening evaluation and according to inclusion/exclusion criteria, they will undergo 3 phases. By randomized crossover design, the subject will receive fexofenadine with water, grapefruit juice, or furanocoumarin-free grapefruit juice.
  Other Names: Screening: labs, physical exam; Placement of an intravenous (IV) line; Collection of blood over 72 hours

SUMMARY:
Purpose: Grapefruit juice is one of the most extensively studied dietary/natural substances shown to interact with a variety of medications. However, unanswered questions remain regarding the causative ingredients and mechanisms underlying such drug-grapefruit juice interactions. Compounds in grapefruit juice called furanocoumarins have been established as major causative ingredients, which act by inhibiting the elimination (metabolism) of drugs, leading to increased circulating drug concentrations. Increased drug concentrations can in turn lead to increased drug potency or even toxicity. Grapefruit juice also has been shown, paradoxically, to decrease circulating concentrations of some drugs, including the non-sedating antihistamine agent, fexofenadine (Allegra), which undergoes negligible metabolism. Whether or not furanocoumarins mediate the decrease in fexofenadine concentrations is unknown. The purpose of the proposed study is to compare the effects of a "furanocoumarin-free" grapefruit juice with grapefruit juice on circulating concentrations of fexofenadine.

DETAILED DESCRIPTION:
Participants: Healthy volunteers of any race/ethnicity, ranging in age from 18 to 65 years, will be enrolled.

Procedures (methods): Procedures will include administration of water, furanocoumarin-free grapefruit juice, or grapefruit juice with fexofenadine; placement of an intravenous (IV) line; and collection of blood over 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 18 and 65
* Normal screening laboratory test results
* Able to understand the informed consent form
* Willing to abstain from grapefruit products and all fruit juices for one week prior to and during the study
* Willing to abstain from alcohol and caffeinated beverages the evening prior to each study day

Exclusion Criteria:

* History of intolerance to grapefruit products
* History of any allergy or hypersensitivity to grapefruit products or fexofenadine
* History of significant medical conditions that the study physician believes would increase risk
* History of significant alcohol abuse and/or illicit drug use
* Tobacco use within the month preceding the study
* Pregnancy or breast-feeding
* Taking concomitant medications, both prescription and non-prescription (including herbal products), known to alter fexofenadine blood levels or P-gp and/or OATP activity (women stabilized on hormonal methods of birth control will be allowed to participate)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Paine, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- North Carolina Clinical and Translational Research Center, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening began in September 2009. Potential eligible subjects presented for a screening visit at the UNC Clinical and Translational Research Center (CTRC) within 1 month prior to the first day of the study.
Pre-assignment Details: No significant events/approaches for overall study following participant enrollment but prior to group assignment. 18 subjects recruited and screened. No exclusions.
Groups:
- Sequence 1: Water, GFJ, Furanocoumarin-free GFJ; Sequence 2: Water, Furanocoumarin-free GFJ, GFJ; Sequence 3: GFJ, Furanocoumarin-free GFJ, Water; Sequence 4: GFJ, Water, Furanocoumarin-free GFJ; Sequence 5: Furanocoumarin-free GFJ, GFJ, Water; Sequence 6: Furanocoumarin-free GFJ, Water, GFJ: By randomized 3-way crossover design, the subject will receive single doses of fexofenadine 120 mg (2 60mg tablets) and 240 mL of water, grapefruit juice (GFJ), and furanocoumarin-free GFJ (depending on Williams design sequence), with at least 10 day washout in between each treatment period.
Period: Period 1 (5 Days)
Arm/Group | Sequence 1: Water, GFJ, Furanocoumarin-free GFJ | Sequence 2: Water, Furanocoumarin-free GFJ, GFJ | Sequence 3: GFJ, Furanocoumarin-free GFJ, Water | Sequence 4: GFJ, Water, Furanocoumarin-free GFJ | Sequence 5: Furanocoumarin-free GFJ, GFJ, Water | Sequence 6: Furanocoumarin-free GFJ, Water, GFJ
Started | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to (and completed) one of six sequences.)
Completed | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1 (10 Days)
Arm/Group | Sequence 1: Water, GFJ, Furanocoumarin-free GFJ | Sequence 2: Water, Furanocoumarin-free GFJ, GFJ | Sequence 3: GFJ, Furanocoumarin-free GFJ, Water | Sequence 4: GFJ, Water, Furanocoumarin-free GFJ | Sequence 5: Furanocoumarin-free GFJ, GFJ, Water | Sequence 6: Furanocoumarin-free GFJ, Water, GFJ
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (5 Days)
Arm/Group | Sequence 1: Water, GFJ, Furanocoumarin-free GFJ | Sequence 2: Water, Furanocoumarin-free GFJ, GFJ | Sequence 3: GFJ, Furanocoumarin-free GFJ, Water | Sequence 4: GFJ, Water, Furanocoumarin-free GFJ | Sequence 5: Furanocoumarin-free GFJ, GFJ, Water | Sequence 6: Furanocoumarin-free GFJ, Water, GFJ
Started | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.)
Completed | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (3-way crossover study. Each subject was his/her own control and underwent all 3 treatments.) | 3 (3-way crossover study. Each subject was his/her own control and underwent all 3 treatments.) | 3 (3-way crossover study. Each subject was his/her own control and underwent all 3 treatments.) | 3 (3-way crossover study. Each subject was his/her own control and underwent all 3 treatments.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2 (10 Days)
Arm/Group | Sequence 1: Water, GFJ, Furanocoumarin-free GFJ | Sequence 2: Water, Furanocoumarin-free GFJ, GFJ | Sequence 3: GFJ, Furanocoumarin-free GFJ, Water | Sequence 4: GFJ, Water, Furanocoumarin-free GFJ | Sequence 5: Furanocoumarin-free GFJ, GFJ, Water | Sequence 6: Furanocoumarin-free GFJ, Water, GFJ
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (5 Days)
Arm/Group | Sequence 1: Water, GFJ, Furanocoumarin-free GFJ | Sequence 2: Water, Furanocoumarin-free GFJ, GFJ | Sequence 3: GFJ, Furanocoumarin-free GFJ, Water | Sequence 4: GFJ, Water, Furanocoumarin-free GFJ | Sequence 5: Furanocoumarin-free GFJ, GFJ, Water | Sequence 6: Furanocoumarin-free GFJ, Water, GFJ
Started | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.) | 3 (3-way crossover study. Each subject was assigned to one of six sequences.)
Completed | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.) | 3 (Each subject served as his/her own control and completed assigned sequence.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Water, GFJ, Furanocoumarin-free GFJ; Sequence 2: Water, Furanocoumarin-free GFJ, GFJ; Sequence 3: GFJ, Furanocoumarin-free GFJ, Water; Sequence 4: GFJ, Water, Furanocoumarin-free GFJ; Sequence 5: Furanocoumarin-free GFJ, GFJ, Water; Sequence 6: Furanocoumarin-free GFJ, Water, GFJ: This randomized, open-label, single-dose, 3-way crossover study in healthy volunteers will be conducted in the CTRC. Once subjects are identified as eligible to participate, based on their screening evaluation and according to inclusion/exclusion criteria, they will undergo 3 phases. By randomized crossover design, the subject will receive fexofenadine with water, grapefruit juice (GFJ), and furanocoumarin-free grapefruit juice (depending on Williams design sequence) with at least 10 day washout in between each treatment period.
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Water, GFJ, Furanocoumarin-free GFJ | Sequence 2: Water, Furanocoumarin-free GFJ, GFJ | Sequence 3: GFJ, Furanocoumarin-free GFJ, Water | Sequence 4: GFJ, Water, Furanocoumarin-free GFJ | Sequence 5: Furanocoumarin-free GFJ, GFJ, Water | Sequence 6: Furanocoumarin-free GFJ, Water, GFJ | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean | 26 (1.0) | 34 (17) | 51 (11) | 39 (11) | 33 (9.1) | 30 (7.5) | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 2 | 1 | 3 | 9
  Male | 1 | 2 | 3 | 1 | 2 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Primary Pharmacokinetic Measure: Area Under the Curve (AUC)
Time Frame: 0-72 hours
Measure: Geometric Mean (Full Range); unit: micromolar*hr
Groups:
- Water; Grapefruit Juice; Furanocoumarin-free Grapefruit Juice: For juice and water comparisons, fexofenadine + grapefruit juice or fexofenadine + furanocoumarin-free grapefruit juice will be the test agent (numerator) and fexofenadine + water will be the reference standard (denominator).
Arm/Group | Water | Grapefruit Juice | Furanocoumarin-free Grapefruit Juice
Number analyzed (Participants) | 18 | 18 | 18
micromolar*hr
  Water | 4.2 [1.7 to 8.4] | 4.2 [1.7 to 8.4] | 4.2 [1.7 to 8.4]
  Grapefruit juice | 3.2 [1.9 to 6.3] | 3.2 [1.9 to 6.3] | 3.2 [1.9 to 6.3]
  Modified grapefruit juice | 3.1 [1.9 to 5.9] | 3.1 [1.9 to 5.9] | 3.1 [1.9 to 5.9]
Statistical Analysis 1: Comparison: Grapefruit Juice vs Furanocoumarin-free Grapefruit Juice; For juice comparisons, fexofenadine + furanocoumarin-free grapefruit juice will be the test agent (numerator) and fexofenadine + grapefruit juice will be the reference standard (denominator); Test type: Superiority or Other; p = 0.78, t-test, 2 sided; Geometric Mean AUC Ratio (GFJ/mGFJ) = 0.96, 90% CI 2-sided [0.4 to 1.5]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sequence 1: Water, GFJ, Furanocoumarin-free GFJ | Sequence 2: Water, Furanocoumarin-free GFJ, GFJ | Sequence 3: GFJ, Furanocoumarin-free GFJ, Water | Sequence 4: GFJ, Water, Furanocoumarin-free GFJ | Sequence 5: Furanocoumarin-free GFJ, GFJ, Water | Sequence 6: Furanocoumarin-free GFJ, Water, GFJ
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No